CLINICAL TRIAL: NCT05988138
Title: Reward Responsiveness as a Prevention Target in Youth At Risk for Anhedonia
Brief Title: Prevention of Anhedonia in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Autumn Kujawa, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 230616
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Anhedonia; Depression
MeSH Terms: conditions — Anhedonia; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Promoting Positive Emotions (Experimental)
  Interventions: Behavioral: Family Promoting Positive Emotions
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Family Promoting Positive Emotions — An 8-week dyadic intervention using cognitive and behavioral skills to up-regulate positive emotions in children and mothers
  Arms: Family Promoting Positive Emotions
Behavioral: Psychoeducation — An 8-week comparison condition that offers education in mental health, depression prevention, and accessing mental health resources
  Arms: Psychoeducation

SUMMARY:
This trial will test the effects of a positive emotion-focused preventive intervention on reward responsiveness in children of mothers with histories of depression and anhedonia.

DETAILED DESCRIPTION:
This study will test the effects of a dyadic preventive intervention, Family Promoting Positive Emotion (F-PPE), for 8- to 12-year-old children of mothers with a history of major depressive disorder (MDD) with anhedonia. The study will first test F-PPE effects on child reward responsiveness (R61), and pending evidence of target engagement, effects on real-world experience of interest/pleasure and clinical symptoms of anhedonia will be evaluated in a second, larger clinical trial (R33). F-PPE was designed to increase child positive valence systems function through mother-child training in behavioral and cognitive skills to increase pleasant activities and attention towards/savoring the positive, individual and dyadic goals, and skills practice. For the R61 phase, eligible child participants (N=60 intervention completers) will complete an EEG assessment of neural reward responsiveness, as well as halfway through the intervention (4 weeks) to determine dose effects. Children and their biological mothers will be randomly assigned to 8 sessions of F-PPE or a psychoeducation comparison condition (groups will be matched on child sex and baseline RewP). Both interventions will be administered through individual telehealth sessions with a masters- or doctoral-level clinician under the supervision of the PIs. To ensure treatment fidelity, videotaped sessions will be reviewed for adherence to the protocol, clinicians will participate in weekly group supervision, and supervisors will randomly review recorded sessions for ratings of treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers with past or current MDD with anhedonia and their 8- to 12-year-old children
* Child and biological mother can read and speak fluently in English
* Child and mother have access to a computer or tablet and internet for videoconferencing
* For compensation purposes, child and biological mothers must be U.S. citizens

Exclusion Criteria:

* Children with past or current major depressive disorder (MDD) and/or anhedonia lasting most of the day, nearly every day for at least 2 weeks based on semi-structured interviews will be excluded
* Mothers or children with intellectual or developmental disabilities
* Mothers with past 6 months substance use disorder with moderate or greater severity
* Children or mothers with a lifetime history of a manic or hypomanic episode/bipolar disorder
* Children or mothers with a psychotic disorder (e.g., schizophrenia)
* Children or mothers with visual or hearing impairments that interfere with completing study measures and sessions
* Child offspring of a mother who has previously participated in the study with another biological child
* Children taking medications for emotional or behavioral problems other than SSRIs (stable dose for 6 weeks before time of enrollment) or psychostimulants

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Neural responses to rewards measured by electroencephalogram (EEG) in a computerized guessing reward task (physiological measure) | 4 and 8 weeks
  The reward positivity (RewP) component will be measured using EEG with an established computerized guessing reward task ("Doors" task). EEG data will be processed using best practices and the RewP component will be exported from the EEG data approximately 250-350 ms after feedback presentation at the electrode Cz. RewP scores will be quantified as the relative neural response to reward vs. loss feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Jesup/Hobbs Building, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Institute of Mental Health Data Archive